CLINICAL TRIAL: NCT05144906
Title: Implicit Attitudes Toward Body Shape Among Blind Women: Evidence From an Auditory Implicit Association Test
Brief Title: Implicit Attitudes Toward Body Shape Among Blind Women
Status: Completed | Type: Observational
Sponsor: University of Haifa (Other)
Responsible Party: Sponsor
Other Study IDs: 493-20
Record Dates: First submitted 2021-11-17; First posted 2021-12-03 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2021-11

CONDITIONS: Blindness; Implicit Bias
MeSH Terms: conditions — Blindness; Bias, Implicit

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Blind women: The blind women group will include women who are congenitally blind or that were blinded early in life (up to the age of 7).
- Sighted women: Women with normal or corrected-to-normal eye sight.

SUMMARY:
High levels of body image concerns and disordered eating in western women have been associated with the promotion of an unrealistically thin body ideal. The pressure to conform with the thin-ideal forms both explicit and implicit attitudes favoring thinness. Visual-based media depicting thin-idealized bodies plays a major role in forming such attitudes. However, attitudes favoring thinness can also be transmitted through non-visual communication such as peer pressure and significant others. The current study will examine if implicit attitudes favoring thinness and disliking overweight bodies can be formed without ever being exposed to visual-based media or being visually exposed to body shapes. To achieve this goal, the study will assess implicit attitudes towards thin and overweight bodies in congenitally blind women and those who were blinded early in life. The assessment will be carried out using a novel auditory weight-bias implicit association test.

DETAILED DESCRIPTION:
Previous studies have demonstrated strong implicit associations between images portraying thin bodies and positive words and images portraying overweight bodies and negative words among healthy individuals in Western society. This so-called "implicit weight bias" is thought to represent individuals' unconscious or automatic stereotypical attitudes against being overweight. The goal of the current study is to examine implicit weight biases among congenitally blind as well as sighted women using a novel auditory version of the weight bias implicit association task. In this task, participants hear a series of words and are requested to classify each word using a motor response to the matching category. The categories used will be negative and positive words as well as words describing thin and overweight bodies. Implicit anti-fat bias is reflected by longer response times and higher error rates, when positive words and those describing overweight bodies require the same motor response and when negative words are coupled with words describing thin bodies compared to when positive and negative words are coupled with words describing thin and overweight bodies, respectively.

The investigators have collected preliminary results in a sample of blind women (N = 18) in Israel. The investigators plan to a) expand the data collection in Israel to reach a sample of 30 blind women and to b) carry out a full replication of the study in an independent sample of blind and sighted women in the US. Data have not been collected yet for the US replication study. Based on the effect size of the the implicit bias effect (represented by the IAT D score) obtained in preliminary results in the Israeli sample (Cohen's D = 0.74), a power analysis using G*power was carried out and showed that a sample of 22 participants is sufficient to detect the IAT implicit bias effect with a power > 95% and an a-priori alpha set at 0.05.

Based on preliminary results in the Israeli sample, it is hypothesized that:

1. Blind women will demonstrate an implicit bias indicating preference for thin bodies and a dislike of overweight bodies. This effect will be reflected by slower response times when words describing thin bodies will be coupled with negative compared to positive words and when words describing overweight bodies will be coupled with positive compared to negative words. This implicit bias effect will be computed using the IAT's D algorithm.
2. The implicit anti-fat bias effect (IAT D-score) will be comparable between sighted and blind women.

ELIGIBILITY:
Blind Women

Inclusion Criteria:

* Aged 18-45 years.
* Congenitally blind or blinded no later than the age of 7.
* Inability to see themselves in the mirror.
* Inability to recognize other people's faces or bodies.
* Inability to use visual-based media.
* Fluent English speakers.

Exclusion Criteria:

• Any condition that prevents the ability to use a computer.

Sighted women

Inclusion Criteria:

* Aged 18-45 years old.
* Corrected or corrected-to-normal vision.
* Fluent English speakers.

Exclusion Criteria:

• Any condition that prevents the ability to use a computer.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The blind women group will only include women who were blinded earlier than the age of 7 and cannot see themselves in the mirror not recognize other people's faces or bodies or use visual-based media. The sighted women group will include women with normal or corrected-to-normal vision.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Implicit Association Test | One assessment at baseline after study information and informed consent was given
  IAT D-Score calculated for assessing an implicit weight bias. The IAT D score will be computed using the improved algorithm suggested by Greenwald et al. (2003). According to this algorithm, RTs longer than 10,000 ms will be deleted. Participants with more than 10% of the trials that are shorted than 300 ms will be excluded from the analysis. Mean RTs for correct trials will be computed for each block separately. Error trials will be replaced by the mean score of each block + 600 ms. Then, the difference in RTs between the practice stereotype incongruent and practice congruent conditions will be divided by their pooled SD. Then, the different in RTs between the test stereotype congruent and incongruent blocks will be divided by their pooled RTs. Lastly, the two scores form the practice and test blocks will be averaged to compute the IAT D score.

SECONDARY OUTCOMES:
Sociocultural Attitudes Toward Appearance Questionnaire-4 (SATAQ-4R) | up to 72 hours after completion of the baseline assessment
  The SATAQ-4R is a gender-specific self-report tool composed of 31 items in the female version. It includes four scales to evaluate the perceived pressure from family, peers, significant others, and the media to attain a thin body and three sub-scales that evaluate the desire to attain a lean body, to attain a muscular physique and overall concern with personal appearance. Participants rate their agreement with various statements on a 5-point scale.
Ideal Body Stereotype Scale-Revised (IBSS-R) | up to 72 hours after completion of the baseline assessment
  The IBSS-R measures the pursuit of the thin beauty ideal. Participants are asked to indicate to what extent they agree with six statements about what attractive women look like on a 5-point scale from strongly disagree to strongly agree. The total sum ranges from 0 to 30 with higher scores indicating a stronger internalization of the thin ideal.
Body Parts Dissatisfaction Scale (BPDS) | up to 72 hours after completion of the baseline assessment
  The BPDS assesses body dissatisfaction by asking the respondents to rate their satisfaction with 9 body parts on a scale from 1 (extremely dissatisfied) to 5 (extremely satisfied). Lower scores represent greater body dissatisfaction.
Body mass index (BMI) | up to 72 hours after completion of the baseline assessment
  Weight and height data will be collected via self-report in order to calculate BMI (kg/cm2).

CONTACTS AND LOCATIONS:
Overall Officials: Noam Weinbach, PhD, Principal Investigator — University of Haifa
Locations (1):
- University of Haifa, Haifa, Central District, Israel

IPD SHARING:
Plan to Share IPD: Yes
The study will provide open access for de-identified data as well as for the analytical plan and protocol.
Supporting Information: Study Protocol, SAP
Time Frame: Upon submission of a manuscript for publication
Access Criteria: Open access